CLINICAL TRIAL: NCT00252928
Title: Health Impact Study of a Water Treatment Tablet, Aquatabs, in Tamale, Ghana
Brief Title: Health Impact Study of Aquatabs in Tamale, Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Medentech (Industry); Emory University Center for Global Safe Water (Other); NewEnergy (Unknown); University for Development Studies, Tamale, Ghana (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: CDC-NCID-4730
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2007-10

CONDITIONS: Diarrhea
Keywords: sodium dichloroisocyanurate; water purification; disinfection; Ghana
MeSH Terms: conditions — Diarrhea | interventions — troclosene; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- A (Placebo Comparator): Placebo group does not receive Aquatabs.
  Interventions: Other: Placebo
- B (Experimental): Intervention arms receives Aquatabs.
  Interventions: Other: Sodium dichloroisocyanurate (NaDCC) tablets

INTERVENTIONS:
Other: Sodium dichloroisocyanurate (NaDCC) tablets — Intervention arm receives NaDCC tablets to use for to disinfect their household water for use for 20L of water. Ideally, disinfection occurs every day.
  Other Names: Aquatabs
  Arms: B
Other: Placebo — Placebo
  Arms: A

SUMMARY:
The purpose of this study to determine whether Aquatabs, a water treatment tablet, reduces diarrheal diseases in a peri-urban population of Tamale, Ghana.

ELIGIBILITY:
Inclusion Criteria:

* Households with at least one child under 5 years old

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2006-07; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Measure the impact of Aquatabs on diarrhea among persons in households in Tamale, Ghana. | 12 weeks

SECONDARY OUTCOMES:
Assess the microbiological quality of household water among persons living in Tamale, Ghana. | 12 weeks
Determine the acceptability of Aquatabs. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seema Jain, MD, Principal Investigator — Centers for Disease Control and Prevention; Robert Quick, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (3):
- Emory University Center for Global Safe Water, Atlanta, Georgia, United States
- Ghana (2):
  - NewEnergy, Tamale
  - University of Development Studies, Tamale

REFERENCES:
- [Background] Mintz ED, Reiff FM, Tauxe RV. Safe water treatment and storage in the home. A practical new strategy to prevent waterborne disease. JAMA. 1995 Mar 22-29;273(12):948-53. PMID 7884954
- [Background] Reiff FM, Roses M, Venczel L, Quick R, Witt VM. Low-cost safe water for the world: a practical interim solution. J Public Health Policy. 1996;17(4):389-408. PMID 9009536
- [Background] Quick RE, Venczel LV, Mintz ED, Soleto L, Aparicio J, Gironaz M, Hutwagner L, Greene K, Bopp C, Maloney K, Chavez D, Sobsey M, Tauxe RV. Diarrhoea prevention in Bolivia through point-of-use water treatment and safe storage: a promising new strategy. Epidemiol Infect. 1999 Feb;122(1):83-90. doi: 10.1017/s0950268898001782. PMID 10098789
- [Background] Quick RE, Venczel LV, Gonzalez O, Mintz ED, Highsmith AK, Espada A, Damiani E, Bean NH, De Hannover EH, Tauxe RV. Narrow-mouthed water storage vessels and in situ chlorination in a Bolivian community: a simple method to improve drinking water quality. Am J Trop Med Hyg. 1996 May;54(5):511-6. doi: 10.4269/ajtmh.1996.54.511. PMID 8644907
- [Background] Sobel J, Mahon B, Mendoza CE, Passaro D, Cano F, Baier K, Racioppi F, Hutwagner L, Mintz E. Reduction of fecal contamination of street-vended beverages in Guatemala by a simple system for water purification and storage, handwashing, and beverage storage. Am J Trop Med Hyg. 1998 Sep;59(3):380-7. doi: 10.4269/ajtmh.1998.59.380. PMID 9749629